CLINICAL TRIAL: NCT05811884
Title: Patient-centered Assessment of the Effects of Powered Exoskeleton Use in People With Spinal Cord Injury
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Financial issues
Sponsor: Istituto Nazionale Assicurazione contro gli Infortuni sul Lavoro (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSC DCAPR Prospettico
Record Dates: First submitted 2023-03-16; First posted 2023-04-13 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- House rehabilitation (Experimental): The subjects will be provided of the powered exoskeleton for home use. No specific indications will be provided, but using the technology as much as possible.
  Every six months, the subjects will be asked to attend a single-day session by the clinical facility (follow-up session) consisting on the assessement of a series of qualitative and quantitative measurements.
  Interventions: Device: Rehabilitation
- Central rehabilitation (Experimental): The subjects will be asked to attend to periodic rehabilitation sessions by the clinical facility. The rehabilitation session will consist in an intense 1-week activities session every three months. Every six months, the subjects will be asked to attend a single-day session by the clinical facility (follow-up session) consisting on the assessement of a series of qualitative and quantitative measurements.
  Interventions: Device: Rehabilitation

INTERVENTIONS:
Device: Rehabilitation — The subjects will be provided of the powered exoskeleton for home use. No specific indications will be provided, but using the technology as much as possible.
  The subjects will be asked to attend to periodic rehabilitation sessions by the clinical facility. The rehabilitation session will consist in an intense 1-week activities session every three months.
  Every six months, the subjects will be asked to attend a single-day session by the clinical facility (follow-up session) consisting on the assessement of a series of qualitative and quantitative measurements.

SUMMARY:
The goal of this clinical trial is to assess the efficacy of the use of powered exoskeleton for ambulation on the quality of life in subjects with spinal cord injury. The main questions it aims to answer are:

1. How much does the use of powered exoskeleton improve the quality of life in subjects with spinal cord injury after a 24 months treatment period in a house context (treatment 1) or in a clinical setting (treatment 2)?
2. How much do the two treatments differ in terms of cost-utility ratio?

Participants will be included in a multi-step process consisting of:

1. Recruitment, based on eligibility criteria;
2. Observation of the "stability" over time (2 months) of specific clinical parameters;
3. Training in the use of the powered exoskeleton (1 month);
4. Random selection of the rehabilitation treatment (house rehabilitation or central rehabilitation); concerning the house rehabilitation, the subject will be provided the device for home use; concerning the central rehabilitation, the subject will be asked to use intensively the device 1-week every three months in a clinical facility.
5. Follow-up: every six months each subject will be asked to attend a single-day activities session consisting of walking activities with the exoskeleton, compilation of questionnaires, sub-maximal effort test with arm-ergometer, and physical examinations made by a physiatrist.

ELIGIBILITY:
Inclusion Criteria:

* Assisted by Inail;
* Age between 18 and 65 years;
* Body weight lower than 113 Kg;
* Level of spinal lesion T4 and higher;
* Integrity of upper limbs (strength and range of motion assessed by a clinical operator);
* Abbreviated Injury Scale (AIS) score A or B;
* Number of months after lesion higher than 6;
* Anthropometry in conformity with the declarations of exoskeleton's manufacturers.

Exclusion Criteria:

* Use of the powered exoskeleton in the last 6 months (in this case a wash-out phase is required);
* Use of colostomy bag;
* The subject is pregnant/ nursing;
* Presence of cognitive impairments;
* Presence of severe neurologic lesions in addition to SCI (sclerosis, cerebral palsy or trauma,…);
* Severe comorbidities;
* Uncontrolled hypertension or orthostatic hypotension;
* Uncontrolled autonomic dysreflexia;
* Problems at the skeletal system: T-score of femoral neck lower than -3 (DEXA examination is required), bone mineral density of proximal tibia or distal femur lower than 0.6 g/cm2, presence of non-recovered fractures, ectopic ossification, unstable spine;
* Kinesiologic impairments of the lower limbs: Ashworth spasticity of hamstrings, quadriceps, gastrocnemius muscles (right/ left) lower than 4, uncontrolled clonic spasm, pathologic contractures: non conformity of the range of motion of ankle/ knee/ hip with the requisites for use of powered exoskeletons for ambulation, presence of pressure lesions, dysmetria: femurs higher than 1.5 cm/ tibias higher than 2 cm;
* Kinesiologic impairments of the upper limbs: limitations at the joints, weakness of shoulder/ elbow/ hand (manual evaluation by a clinician), no autonomy in transfers;
* Weak control of the trunk;
* Inability to stand for at least 30 minutes;
* Presence of joint prostheses in upper and lower limbs;
* Use of drugs that may affect cognition and coordination while using the exoskeleton.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-10 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life (QoL) | This outcome will be assessed at the baseline and immediately after the intervention
  Short Form-36 questionnaire (SF-36): Generic health status measure. It applies to all health conditions and contains 36 items, divided in 8 domains. The higher the score, the higher the QoL.

SECONDARY OUTCOMES:
Incremental cost utility ratio (ICUR) associated to the treatment | This outcome will be assessed immediately after the intervention
  Incremental cost utility ratio (ICUR) associated to the treatment: it provides healthcare decision- makers and providers with a straightforward information, that is, how much a "unit of utility improvement" would cost them and/or the society. Assuming a timeframe of analysis and two alternative technologies or treatments A and B, ICUR is the ratio between the difference in costs and the difference in utility of A and B
Incidence of Treatment-Emergent Adverse Events assessed by self-report and extracted from the medical records | This outcome will be assessed immediately after the intervention
  Incidence of major adverse events related to the exoskeleton use: falls, bone fractures, skin lesions, pressure lesions, cardiovascular events
Active use assessed by the number of strides and steps performed with the exoskeleton. | This outcome will be assessed immediately after the intervention.
  Strides and steps performed with the exoskeleton are counted automatically by the exoskeleton system. This parameters can be monitored by connecting to the exoskeleton system via a proprietary software.
Change in usability assessed by the System Usability Scale (SUS) questionnaire | This outcome will be assessed at the baseline and at the months 6, 12, 18, 24
  The SUS evaluates the usability of the assistive technology. It consists in 10 items with five response options for respondents, from Strongly agree to Strongly disagree. The participant's scores for each question are converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. The higher the score, the higher the usability.
Change in satisfaction assessed by the Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST) questionnaire | This outcome will be assessed at the baseline and at the months 6, 12, 18, 24
  The QUEST evaluates a person's satisfaction with the assistive technology. It yields three scores: (i) Device, (ii) Services, and (iii) a total QUEST score. (i) consists of 10 items with five response options for respondents, from Strongly agree to Strongly disagree; the score is calculated by averaging the valid item responses; score range: 1-5. (ii) consists of 4 items with five response options for respondents, from Strongly agree to Strongly disagreeare; the score is calculated by averaging the valid item responses; score range: 1-5. (iii) is calculated by averaging the score of (i) and (ii). The QUEST presents a final section where the participants must indicate the three most important features of the technology.
Change in mental status assessed by the Patient Health Questionnaire-9 (PHQ-9) questionnaire | This outcome will be assessed at the baseline and at the months 6, 12, 18, 24
  The PHQ-9 aims at identifying probable major depressive disorder among adult primary care patients. It consists in 9 items with four response options for respondents, from Never to Almost always. The final score is calculated by summing the valid item responses. Score range: 0 -27. The higher the score, the higher the level of depression.
Change in mental status assessed by the General Anxiety Disorder Scale (GAD-7) questionnaire | This outcome will be assessed at the baseline and at the months 6, 12, 18, 24
  The GAD-7 assesses participant's anxiety. It consists of 7 items with four response options for respondents, from Never to Almost always. The final score is calculated by summing the valid item responses. Score range: 0 -21. The higher the score, the higher the level of anxiety.
Change in fitness level assessed by the Metabolic Equivalents of Tasks (METs) associated to the consumption of oxygen (VO2) during a sub-maximal arm crank ergometer test | This outcome will be assessed at the baseline and at the months 6, 12, 18, 24
  The VO2 consumption is measured with a metabolic system throughout an exercise protocol with an arm-ergometer. According to previous study protocols, the VO2 consumption in the last 30 seconds of the arm-ergometer test are used to estimate the peak of VO2 consumption. After, this value is converted in METs.
Change in muscular spasticity assessed by the Modified Ashworth Scale (MAS) | This outcome will be assessed at the baseline and at the months 6, 12, 18, 24
  The MAS assesses the resistance to passive range of motion about a single joint with a 6-point rating scale. It's performed by extending the patients limb first from a position of maximal possible flexion to maximal possible extension ( the point at which the first soft resistance is met). Afterwards, the modified Ashworth scale is assessed while moving from extension to flexion. The higher the score, the higher the muscular spasticity. The scores can assume the following values: 0 - No increase in tone;1 - slight increase in tone giving a catch when slight increase in muscle tone, manifested by the limb was moved in flexion or extension; 1+ - slight increase in muscle tone, manifested by a catch followed by minimal resistance throughout the range of motion; 2 -more marked increase in tone but more marked increased in muscle tone through most limb easily flexed; 3 - considerable increase in tone, passive movement difficult; 4 - limb rigid in flexion or extension.
Change in integrity of the rotator cuff muscles assessed by Jobe's test and Speed's test | This outcome will be assessed at the baseline and at the months 6, 12, 18, 24
  The Jobe's test aids in diagnosing rotator cuff tears or subacromial impingement. The examiner passively elevates the patient's shoulder to 90 degrees of abduction with internal rotation. The examiner then applies a downward pressure against the arm. A positive test is the provocation of pain or abnormal weakness.
  The Speed's test is used to test for superior labral tears or bicipital tendonitis. To perform the Speed's Test, the examiner places the patient's arm in shoulder flexion, external rotation, full elbow extension, and forearm supination; manual resistance is then applied by the examiner in a downward direction. The test is considered to be positive if pain in the bicipital tendon or bicipital groove is reproduced In both test, the exerted force will be also measured using a dynamometer.
Change in self-care and independence assessed by the Spinal Cord Independence Measure (SCIM) questionnaire | This outcome will be assessed at the baseline and at the months 6, 12, 18, 24
  The SCIM assesses of the ability of SCI patients to perform basic activities of daily living. It assesses three subscales: (i) self-care, (ii) respiration and sphincter management, and (iii) mobility. (i) consists in 6 items with four or five response options for respondents. Score range: 0-20. (ii) consists in 4 items with three to six response options for respondents. Score range: 0-40. (iii) consists in 8 items with three to nine response options for respondents. Score range: 0-40. Each subscale score is evaluated separately by summing the valid item responses. The higher the score, the higher the level of independence.
Change in pain assessed by Visual Analogue Scale (VAS) | This outcome will be assessed at the baseline and at the months 6, 12, 18, 24
  The pain VAS is a unidimensional measure of pain intensity, used to record patients' pain progression. It consists in a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (pain in this case) orientated from the left (worst) to the right (best).
Change in sphincter's functionality assessed by a 5-Likert scale | This outcome will be assessed at the beginning of the trial and at each follow-up (every 6 months) until trial completion
  The 5-Likert scale consists of a single item which investigates the patients self-perceived sphincter's functionality, ranging from 1 (worst case) to 5 (best case)
Change in velocity during ambulation assessed by the 6 Minutes Walking Test (6 MWT) | This outcome will be assessed at the baseline and at the months 6, 12, 18, 24
  The 6 MWT is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Change in velocity during ambulation assessed by the 10 Meters Walking Test (10 MWT) | This outcome will be assessed at the baseline and at the months 6, 12, 18, 24
  The 10 MWT is a performance measure used to assess walking speed in meters per second over a short distance. It can be employed to determine functional mobility, gait, and vestibular function.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Protesi Inail, Budrio, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No
Pseudonymized data could be shared upon request only